CLINICAL TRIAL: NCT06135233
Title: Implementation and Outcome of Minimally Invasive Pancreatoduodenectomy in Europe: A Critical Appraisal of the First 3 Years of the E-MIPS Registry
Brief Title: Implementation and Outcome of Minimally Invasive Pancreatoduodenectomy in Europe:
Acronym: E-MIPS
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.G. Besselink, professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NP5626
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pancreas Disease
Keywords: registry; minimally invasive surgery; robot-assisted; laparoscopy; pancreatoduodenectomy; pancreatic surgery
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — all patients undergoing minimally invasive pancreatic surgery, no intervention, no randomization

SUMMARY:
A planned analysis of outcomes among consecutive patients after MIPD from centers participating in the E-MIPS registry (2019-2021). Main outcomes of interest were major morbidity (Clavien-Dindo grade ≥3) and 30-day/in-hospital mortality.

DETAILED DESCRIPTION:
The European registry for Minimally Invasive Pancreatic Surgery (E-MIPS) is an E-AHPBA endorsed registry with the aim to monitor and safeguard the introduction of MIPD in Europe. International multicenter audit-based studies focusing on outcomes of minimally invasive pancreatoduodenectomy (MIPD) are lacking.

A planned analysis of outcomes among consecutive patients after MIPD from centers participating in the E-MIPS registry (2019-2021). Main outcomes of interest were major morbidity (Clavien-Dindo grade ≥3) and 30-day/in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

- Data from all patients who underwent R-MIPD and L-MIPD between January 1st 2019 and December 31st 2021 were included

Exclusion Criteria:

* Other pancreatic procedures
* Hybrid approaches (reconstruction phase open)
* Procedures with insufficient baseline data / missing primary outcome data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from all patients who underwent R-MIPD and L-MIPD between January 1st 2019 and December 31st 2021 were included
Sampling Method: Non-Probability Sample
Enrollment: 1336 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Major morbidity | 30 days
30-day/in-hospital mortality. | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, locatie AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No